CLINICAL TRIAL: NCT07178847
Title: Evaluation of Circulating DNA as a Biomarker of Residual Disease After Chemoradiotherapy for Locally Advanced Head and Necksquamous Cell Carcinoma
Brief Title: cDNA and Residual Disease After Chemoradiotherapy for Locally Advanced Head and Neck Squamous Cell Carcinomas
Acronym: NeckTAR-IN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2025-A01108-41
Record Dates: First submitted 2025-09-03; First posted 2025-09-17 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Head and Neck Carcinoma
Keywords: circulating DNA; residual disease
MeSH Terms: conditions — Neoplasm, Residual | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: All the patients will have a blood sample collected one month after the end of chemoradiotherapy and another at three months (excepted if already done in the main study NeckTAR, e.g., if patient have residual disease and an indication for salvage adenectomy).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cDNA detection (Experimental)
  Interventions: Biological: blood sampling

INTERVENTIONS:
Biological: blood sampling — The intervention consist in blood samples (18mL) collected 1 and 3-months after the end of chemoradiotherapy

SUMMARY:
The goal of this ancillary clinical trial is to evaluated circulating DNA as a biomarker of residual disease after chemoradiotherapy for locally advanced head and neck squamous cell carninoma.

The main question it aims to answer is :

- Does circulating DNA (cDNA) be able to detect residual disease 3 months after the end of chemoradiotherapy ? Researchers will compare detection of cDNA at 3-months and objective response (clinical and radiological).

Participants will :

* be included in the main study (Neck-TAR)
* have a blood sample 1 and 3-month after the end of treatment

ELIGIBILITY:
Selection Criteria:

* Patient included in NeckTAR study
* Written informed consent signed for NeckTAR-IN study
* Affiliation to the French social security system

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
cDNA detection and objective response 3 months after the end of chemoradiotherapy | 3 months after chemoradiotherapy
  The detection or non detection of cDNA after treatment will be compared with the objective response (complete response versus progression/stability/partial response)

SECONDARY OUTCOMES:
cDNA detection and objective response one month after the end of chemoradiotherapy | 1 month after the end of chemoradiotherapy
  The detection or non detection of cDNA after treatment will be compared with the objective response (complete response versus progression/stability/partial response)
Overall survival | At the end of the main study (27 months after the end of treatment)
  The overall survival is defined as the time between the date of inclusion and the date of death from any cause.
Progression-free survival | At the end of the main study (27 months after the end of treatment)
  The progression-free survival is defined as the time between the date of inclusion and the date of the first progression of the disease (clinical or radiological) or death from any cause.
cDNA kinetic | 1- and 3-month after the end of chemoradiotherapy
  cDNA detection at 1 and 3 months after the end of chemoradiotherapy
Concordance of mutational profiles and HPV-HR genotypes between primary tumor, ctDNA at diagnosis and ctDNA | 1- and 3-months after the end of chemoradiotherapy
  This will be evaluated according to the mutational profile determined by NGS at each timepoint
Determining the most frequent mutations. | 3-months after the end of chemoradiotherapy
  That will be evaluated by analysing the results of NGS (among the 194 genes in our panel)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen BERNADACH Coordinator, MD, Study Director — Centre Jean Perrin
Locations (3):
- France (3):
  - Centre Jean PERRIN, Clermont-Ferrand, Puy-de-Dôme
  - Hôpital de la Croix-Rousse, Lyon
  - CHU de Saint-Étienne, Saint-Etienne